CLINICAL TRIAL: NCT01442623
Title: Conventional Versus Virtual Reality Based Vestibular Rehabilitation; Effect on Dizziness, Gait and Balance
Brief Title: Conventional Versus Virtual Reality Based Vestibular Rehabilitation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Beaumont Hospital (Other); Emory University (Other); Royal Victoria Eye and Ear Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RoyalCSI DMeldrum
Record Dates: First submitted 2011-09-21; First posted 2011-09-28 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Peripheral Vestibular Disease
Keywords: Vestibular Rehabilitation; Balance; Virtual Reality; Gait; Dizziness
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Vestibular Rehabilitation (Active Comparator): Six week program of conventional vestibular rehabilitation.
  Interventions: Other: Vestibular Rehabilitation
- Nintendo Wii Vestibular Rehabilitation (Experimental): Six week program of vestibular rehabilitation using the Nintendo Wii Fit Plus.
  Interventions: Other: Vestibular Rehabilitation

INTERVENTIONS:
Other: Vestibular Rehabilitation — The patients in the Nintendo Wii Vestibular Rehabilitation group will undergo a standardised 6 week program of vestibular rehabilitation using the Nintendo Wii Fit Plus at home 5 times a week. They will perform a series of exercises and games on the Wii Fit Plus that are designed to challenge and retrain balance. They will be seen once a week by a physiotherapist for review and progression of exercises.
  Patients in the Conventional Vestibular Rehabilitation group will undergo a standardised program of conventional vestibular rehabilitation using conventional balance exercises (Herdman 2007) 5 times a week. They will be seen once a week by a physiotherapist to progress exercises and will receive a standardised home exercise program.
  Other Names: Balance retraining; Virtual reality rehabilitation

SUMMARY:
Dizziness is a common and disabling symptom and is associated with unsteadiness in both standing and walking, sometimes resulting in falls. People who have any of these problems often have a disease process affecting the inner ear. A proportion of people will recover spontaneously over time; those that do not may benefit from a specialized form of physiotherapy known as vestibular rehabilitation. This consists of exercise regimes that are individualized to each person depending on their problems. These regimes aim to decrease dizziness, help patients to re-learn movement patterns and improve their balance during standing and walking. There is considerable research supporting vestibular rehabilitation but it is not clear what is the best type, setting or frequency of treatment. How therapy impacts on walking ability is also not clear. Recent developments have suggested that force plate and virtual reality therapies may benefit. This form of therapy can provide feedback that is unavailable with conventional exercises. Exposure to virtual environments can challenge balance which helps to retrain it. The aim of this study is to compare conventional vestibular rehabilitation with a force plate/virtual reality therapy based vestibular rehabilitation, using a universally available virtual reality system (Nintendo Wii Fit Plus®). In this study, consenting patients with a vestibular disorder will be assigned randomly to either a conventional treatment or a virtual reality based treatment that is customized to their individual problems. They will receive treatment for 8 weeks. The effects of treatment will be measured by state of the art computerized analysis of walking and balance. Questionnaires that obtain information about how severe their dizziness is will also be administered. The study will help therapists understand how inner ear problems affect walking and balance. It will also provide information on the optimum method of providing vestibular rehabilitation and thus improve patient care.

DETAILED DESCRIPTION:
Unilateral vestibular disease results in vertigo, dizziness, dysequilibrium and gait problems. Recovery results from a process known as vestibular compensation where visual and proprioceptive inputs are upregulated, or remaining vestibular function is recalibrated and utilised more effectively (Curthoys, 2000). Patients who do not compensate remain significantly impaired. They benefit from specialised assessment and treatment techniques collectively referred to as vestibular rehabilitation (Hillier and McDonnell, 2011). This form of rehabilitation has its roots in the empirical work of Cawthorne and Cooksey, who in the 1940's first documented the important role of exercise in recovery after a vestibular injury (Cooksey, 1945) and more recently in studies investigating vestibular adaptation (Schubert et al., 2008). Vestibular rehabilitation programs can be considered as motor learning programs and thus require practice and feedback. In conventional rehabilitation it is difficult for patients to gain feedback of performance performing balance exercise which can be repetitive and boring. Force plate technology has been used in the clinical setting to provide visual and auditory feedback and has shown some promising results (Teggi et al., 2009). Virtual reality, defined as 'a high-end-computer interface that involves real time simulation and interactions through multiple sensorial channels' (Burdea and Coiffet, 2003) is also being investigated in laboratory settings. There is some support for the use of virtual reality in vestibular rehabilitation (Viirre and Sitarz, 2002) but these technologies are presently prohibitively expensive and are not universally available. They require considerable therapist time and are unlikely to be used with the frequency that is required for motor learning (particularly in vestibular rehabilitation where most programs entail daily exercise). Recent developments in the gaming industry have resulted in the Nintendo Wii ® Fit Plus, which combines a force platform with an accelerometer to provide visual and auditory feedback of subjects' centre of gravity during virtual reality exercises and games. It stimulates movement and perturbs balance in order to retrain it. Use of this low cost gaming system could easily be adapted to meet the requirements of a vestibular rehabilitation program. The system allows for accurate monitoring of use in terms of time and frequency which is an area that has proven difficult to monitor in both research and clinical applications due to inaccurate patient recall. It is fun to use and therefore may be motivating patients. The rehabilitation community is beginning to investigate this technology in the area of balance retraining (Nitz et al. 2009). Anecdotal reports indicate the Wii is being used in vestibular rehabilitation (Hain, 2011) but as yet no randomised controlled trials exist.

It is important to measure the effect of this technology which can easily be incorporated into the home environment and compare it to conventional treatment before it can be recommended for use. In tandem with this is also important to gain some insights into patient satisfaction with both treatments.

Aim To compare the outcome from conventional vestibular rehabilitation to virtual reality based vestibular rehabilitation in the treatment of unilateral vestibular disease.

Objectives To compare the effect of conventional vestibular rehabilitation and virtual reality based rehabilitation on gait.

To compare the effect of conventional vestibular rehabilitation and virtual reality based rehabilitation on subjective complaints of dizziness/vertigo.

To compare the effect of conventional vestibular rehabilitation and virtual reality based rehabilitation on balance.

To compare the effect of conventional vestibular rehabilitation and virtual reality based vestibular rehabilitation on dynamic visual acuity.

To quantify patient satisfaction with conventional and virtual reality based vestibular rehabilitation.

Trial design

The study design will be an assessor blinded randomised controlled trial. There is moderate to strong evidence in the literature for the efficacy of vestibular rehabilitation, therefore a "no" treatment group is not deemed ethical.

Participants

Patients attending the otolaryngology and neurology outpatient clinics in Beaumont Hospital or the Royal Victoria Eye and Ear Hospital will be invited to participate in the trial.

Sample Size Calculation.

Allowing for a 10% drop out, a maximum of 48 participants will need to be recruited for each group (at 80% power to detect p<0.05 on all outcomes). A two year recruitment period is required.

The inclusion criteria will be;

* Clinical diagnosis of peripheral vestibular dysfunction and no other neurological deficit (confirmed where possible with vestibular function testing; canal paresis >20%).
* One of the following subjective complaints indicating a failure of vestibular compensation; disequilibrium, gait instability, vertigo/dizziness, motion sensitivity.
* Not taking medication for vertigo or willing to discontinue with permission from consultant physician.

The exclusion criteria will be;

* Bilateral peripheral vestibular pathology.
* CNS involvement.
* Fluctuating Symptoms (Meniere's disease, migrainous vertigo) or active BPPV.
* Other medical conditions in the acute phase (orthopaedic injury).
* Previous vestibular rehabilitation.
* Pacemaker, Epilepsy (as per Nintendo Wii Guidelines).
* Unwilling or unable to use a Nintendo Wii.

Randomisation

Following baseline assessments participants will be randomised to one of two groups;

1. Conventional vestibular rehabilitation
2. Virtual reality vestibular rehabilitation A third party (not involved in the day to day running of the trial) will use an online randomisation program to assign participants to either conventional treatment or virtual reality treatment in advance of recruitment. The treating physiotherapist will be informed of group allocation after consent has been obtained and after baseline assessments are completed.

Intervention

Based on current evidence in the literature a time frame of up to 6 treatments over 8 weeks will be provided. The interventions for both groups are based on six identified core elements of vestibular rehabilitation used in current clinical practice- education, relaxation, adaptation exercises, habituation exercises, balance and gait retraining and re-conditioning (Meldrum and McConn Walsh, 2011). Programs will be customised to each participant depending on their presenting symptoms and impairments, and will be progressive. All participants will be asked to perform a home exercise program daily for 30 minutes. Where participants are deemed at risk of falling, they will be provided with the necessary preventative instructions. Participants in the virtual reality group will be instructed in the use of the Nintendo Wii ® and will be given one on loan. They will be provided with a customised program which is the virtual reality equivalent of conventional exercises. Those in the conventional group will be provided with a foam balance mat. Participants will be seen weekly for re-assessment, progression of exercises and advice.

Measurement of compliance with home treatment

All participants will be provided with a diary to record compliance with the home exercise program. The Nintendo Wii ® fit plus records type, duration and frequency of exercises and this will also be used as the record for the virtual reality group.

Data will be entered and coded in Microsoft Excel and statistical analysis will be performed using PASW and Stata 11. Intention to treat analysis will be performed. Data will be examined for normality and if a normal distribution is observed t-tests, and an ANOVA model will be used for analysis of interval data with an adjustment for baseline values. The non-parametric equivalent will be used where data are not normally distributed or are non-parametric. Differences from baseline will be calculated for primary and secondary outcomes within groups and between groups at each time point. A significance level of p<0.05 will be set. Effect sizes for within and between groups comparison will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of peripheral vestibular dysfunction and no other neurological deficit (confirmed where possible with vestibular function testing; canal paresis >20%).
* One of the following subjective complaints indicating a failure of vestibular compensation; disequilibrium, gait instability, vertigo/dizziness, motion sensitivity.
* Not taking medication for vertigo or willing to discontinue with permission from consultant physician.

Exclusion Criteria:

* Bilateral peripheral vestibular pathology.
* CNS involvement.
* Fluctuating Symptoms (Meniere's disease, migrainous vertigo) or active BPPV.
* Other medical conditions in the acute phase (orthopaedic injury).
* Previous vestibular rehabilitation.
* Pacemaker, Epilepsy (as per Nintendo Wii Guidelines).
* Unwilling or unable to use a Nintendo Wii.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-02; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Gait Speed (metres per second) | 8 weeks
  Gait speed will be measured using a 5-camera Vicon™ computerised three dimensional gait analysis system.

SECONDARY OUTCOMES:
Computerised Dynamic Posturography | 8 weeks
  Balance will be assessed using computerised dynamic posturography (Equitest, Neurocom).
Vestibular Rehabilitation Benefit Questionnaire | 8 weeks
  The Vestibular Rehabilitation Benefit Questionnaire (Morris et al 2008,2009) is a validated 22 item, 3 part questionnaire that allows participants to rate their dizziness and how it is affecting their quality of life. Clinically meaningful change has been established on the subscores and total scores on this questionnaire.
Hospital Anxiety and Depression Score | 8 weeks
  The Hospital Anxiety and Depression Scale (Zigmond and Snaith, 1983) is a validated scale that has been used previously in studies in vestibular rehabilitation and assesses non-somatic symptoms of anxiety and depression. Scores range between 0 and 21 on each subscale, scores between 8 and 10 are considered borderline and those above ten indicate clinical depression or anxiety
Dynamic Visual Acuity | 8 weeks
  Dynamic visual acuity (DVA) is a measure of how clearly participants can see as their head is moving (a role of the vestibular system). DVA will be measured using Micromedical's™ DVA system of head horizontal plance rotations of 50/100/150 degrees per second and will be compared to static visual acuity.
Activities Balance Confidence Questionnaire | 8 weeks
  The Activities Balance Confidence Questionnaire (Parry et al 2001) is a 16 item questionnaire which asks a participant to rate their balance confidence on a range of activities of daily living.
Patient Satisfaction | 8 weeks
  This is a 15 item questionnaire which asks a participant to rate their satisfaction with the treatment program they underwent in the study, addressing difficulty, motivation, compliance, tiredness after exercise,and enjoyment of the program.

CONTACTS AND LOCATIONS:
Overall Officials: Dara Meldrum, MSc., Principal Investigator — Royal College of Surgeons in Ireland; Susan J Herdman, PhD, Study Director — Emory University; Rory McConn-Walsh, MD, Study Director — Royal College of Surgeons in Ireland
Locations (2):
- Ireland (2):
  - Beaumont Hospital, Dublin, Co. Dublin
  - Royal Victoria Eye and Ear Hospital, Dublin

REFERENCES:
- [Background] Curthoys IS. Vestibular compensation and substitution. Curr Opin Neurol. 2000 Feb;13(1):27-30. doi: 10.1097/00019052-200002000-00006. PMID 10719646
- [Background] Hillier SL, McDonnell M. Vestibular rehabilitation for unilateral peripheral vestibular dysfunction. Clin Otolaryngol. 2011 Jun;36(3):248-9. doi: 10.1111/j.1749-4486.2011.02309.x. No abstract available. PMID 21752206
- [Background] Schubert MC, Migliaccio AA, Clendaniel RA, Allak A, Carey JP. Mechanism of dynamic visual acuity recovery with vestibular rehabilitation. Arch Phys Med Rehabil. 2008 Mar;89(3):500-7. doi: 10.1016/j.apmr.2007.11.010. PMID 18295629
- [Background] Morris AE, Lutman ME, Yardley L. Measuring outcome from Vestibular Rehabilitation, Part I: Qualitative development of a new self-report measure. Int J Audiol. 2008 Apr;47(4):169-77. doi: 10.1080/14992020701843129. PMID 18389412
- [Background] Morris AE, Lutman ME, Yardley L. Measuring outcome from vestibular rehabilitation, part II: refinement and validation of a new self-report measure. Int J Audiol. 2009 Jan;48(1):24-37. doi: 10.1080/14992020802314905. PMID 19173111
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Parry SW, Steen N, Galloway SR, Kenny RA, Bond J. Falls and confidence related quality of life outcome measures in an older British cohort. Postgrad Med J. 2001 Feb;77(904):103-8. doi: 10.1136/pmj.77.904.103. PMID 11161077
- [Background] Teggi R, Caldirola D, Fabiano B, Recanati P, Bussi M. Rehabilitation after acute vestibular disorders. J Laryngol Otol. 2009 Apr;123(4):397-402. doi: 10.1017/S0022215108002983. Epub 2008 Jun 13. PMID 18549515
- [Background] Meldrum D, McConn Walsh R. Vestibular Rehabilitatin IN: Stokes M, Stack E. Physical management in neurological rehabilitation. 3rd ed. Edinburgh: Elsevier; 2011.
- [Background] Viirre E, Sitarz R. Vestibular rehabilitation using visual displays: preliminary study. Laryngoscope. 2002 Mar;112(3):500-3. doi: 10.1097/00005537-200203000-00017. PMID 12148861
- [Background] Cooksey FS. Rehabilitation in Vestibular Injuries. Proc R Soc Med. 1946 Mar;39(5):273-8. doi: 10.1177/003591574603900523. No abstract available. PMID 19993269
- [Background] Nitz JC, Kuys S, Isles R, Fu S. Is the Wii Fit a new-generation tool for improving balance, health and well-being? A pilot study. Climacteric. 2010 Oct;13(5):487-91. doi: 10.3109/13697130903395193. PMID 19905991
- [Background] Herdman S. Vestibular rehabilitation. 3rd ed. Philadelphia: F.A. Davis; 2007.
- [Background] Burdea, G. & Coiffet, P. (2003) Virtual Reality Technology, New Jersey, Wiley and Sons.
- [Derived] Meldrum D, Herdman S, Vance R, Murray D, Malone K, Duffy D, Glennon A, McConn-Walsh R. Effectiveness of conventional versus virtual reality-based balance exercises in vestibular rehabilitation for unilateral peripheral vestibular loss: results of a randomized controlled trial. Arch Phys Med Rehabil. 2015 Jul;96(7):1319-1328.e1. doi: 10.1016/j.apmr.2015.02.032. Epub 2015 Apr 2. PMID 25842051
- [Derived] Meldrum D, Herdman S, Moloney R, Murray D, Duffy D, Malone K, French H, Hone S, Conroy R, McConn-Walsh R. Effectiveness of conventional versus virtual reality based vestibular rehabilitation in the treatment of dizziness, gait and balance impairment in adults with unilateral peripheral vestibular loss: a randomised controlled trial. BMC Ear Nose Throat Disord. 2012 Mar 26;12:3. doi: 10.1186/1472-6815-12-3. PMID 22449224
- See also: Hain T ( Accessed 2011) — http://www.dizziness-and-balance.com